CLINICAL TRIAL: NCT03566251
Title: The Investigation of the Relationship Between Core Stability and Trunk Position Sense With Balance and Functional Mobility in Patients With Multiple Sclerosis
Brief Title: Core Stability, Trunk Position Sense, Balance and Functional Mobility in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 228
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Physical Therapy
Keywords: Multiple Sclerosis; Balance; Core Stability; Proprioception; Functional Mobility
MeSH Terms: conditions — Multiple Sclerosis | interventions — Core Stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Sclerosis (Experimental): Patients with confirmed diagnosis of clinically definite MS, Expanded Sisability Status Scale range of 0.5-4 who are able to walk independently.
  Interventions: Other: Balance; Other: Functional mobility; Other: Core stability; Other: Trunk position sense
- Healthy individuals (No Intervention): 29 healthy volunteers with matching ages and genders

INTERVENTIONS:
Other: Balance — Balance was assessed by Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). Postural Stability (PS), Limits of Stability (LOS) and Modified Sensory Organization Tests (MSOT) were evaluated with this system. PS test assesses static balance during standing up by the ability to hold the center of gravity on the support surface. The test was performed on both feet and on the left and right foot separately. LOS test assesses how much the center of gravity is displaced on the support surface without losing balance during the standing position. MSOT assesses the effects of somatosensory, visual and vestibular senses on postural control during the standing position. It evaluates the sensory component of balance in two different visual conditions and on two different support surfaces.
  Arms: Multiple Sclerosis
Other: Functional mobility — Timed Up and Go (TUG) tests were used to evaluate functional mobility. The TUG measures the time it takes a subject to stand up from an armchair, walk a distance of 3 m, turn, walk back to the chair and sit down. Time was recorded in seconds with a stopwatch.
  Arms: Multiple Sclerosis
Other: Core stability — Core endurance and core strength, which are two specific components of core stability, were evaluated separately. Trunk flexor, trunk extensor, right and left side bridge and prone bridge tests were applied to assess the endurance of the core muscles. Tests were terminated when the subjects said they could not continue the test or when the test position was broken. A stopwatch was used for the measurements and the results were recorded in seconds. The power of core muscles was evaluated with sit-ups and modified push-ups tests. It was recorded how many times the subject could do each test for 30 seconds. The tests were repeated twice and the best measurement score was recorded for use in the statistical analyses.
  Arms: Multiple Sclerosis
Other: Trunk position sense — Trunk position sense was evaluated by the trunk reposition test with Dualer IQ digital inclinometer (J-TECH medical, Salt Lake City, UK, USA). Measurements were made in two levels: lumbosacral (LS) and thoracosacral (TS) regions. The testing took place while standing under three visual-surface conditions. Participants flexed the trunk approximately 30° in the sagittal plane, holding the position for a count of 3 seconds (position 1) and then participants attempted to repeat the previously attained angle. Participants indicated verbally when they felt they had reached the angle and held their position for a count of 3 seconds (position 2). The absolute difference in degrees between positions 1 and 2 was defined as the trunk reposition error (TRE) degree. Participants generated five scores for each visual-surface condition. For each condition, the highest and lowest scores were discarded and the mean of the remaining three scores represented the TRE score
  Arms: Multiple Sclerosis

SUMMARY:
The aim of this study is to compare balance, functional mobility, core stability and trunk position sense in patients with Multiple Sclerosis (PwMS) and healthy controls and investigate the relationship between core stability and trunk position sense with balance and functional mobility in PwMS.

Balance and mobility disorders are seen in various degrees in patients with Multiple Sclerosis (PwMS). Balance and mobility impairments are observed in the beginning with the early period and are one of the most common causes of disability in PwMS.

Coordination between the peripheral sensory system, the central sensory-motor system and the musculoskeletal system which generates motor responses is required to provide balance. If one or more of these systems do not function properly, this results in deficiency in trunk stability and also causes balance and mobility disorders.

It has been shown that balance and mobility disorders are mostly associated with loss of strength, spasticity, coordination disorders and sensory loss. Especially, it is known that strength of core are related to balance and mobility. Although core muscle strength is a significant element of trunk stability, position sense is also responsible for trunk stability. When literature is examined, there is no study which examines the relationship between balance and mobility with core muscles' strength and trunk position sense in PwMS. For all these reasons, we think that balance and functional mobility may be related to core stability and trunk position sense in PwMS

DETAILED DESCRIPTION:
Our study was carried out with the purpose of comparing balance, functional mobility, core stability and trunk position sense in PwMS and healthy controls and investigating the relationship between core stability and trunk position sense with balance and functional mobility in PwMS.

45 PwMS and 29 healthy volunteers with matching ages and genders were included the study. Balance was assessed by Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). Timed Up and Go (TUG) tests were used to evaluate functional mobility. Core endurance and core strength, which are two specific components of core stability, were evaluated separately. Trunk flexor, trunk extensor, right and left side bridge and prone bridge tests were applied to assess the endurance of the core muscles. The power of core muscles was evaluated with sit-ups and modified push-ups tests. Trunk position sense was evaluated by the trunk reposition test with Dualer IQ digital inclinometer (J-TECH medical, Salt Lake City, UK, USA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Sclerosis Disease
* Must be able to walk independently
* The level of disability should be between 0.5-4 according to EDSS

Exclusion Criteria:

* Having acute attack (three months prior to the study)
* Having vision and circulatory system problems,
* Orthopedic problems and pain in the spine, hip, knee or ankle
* Mini-Mental State Examination Test score of less than 25 points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Balance | 1 month
  Balance was assessed by Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). Postural Stability was evaluated with this system (Biodex Medical Systems, 2009). Postural Stability test was performed on both feet and on the left and right foot separately. Total stability index score was obtained as the test result.
Balance | 1 month
  Balance was assessed by Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). Limits of Stability was evaluated with this system (Biodex Medical Systems, 2009). Limits of Stability test assesses how much the center of gravity is displaced on the support surface without losing balance during the standing position. Total direction control score was obtained as the test result.
Balance | 1 month
  Balance was assessed by Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). Modified Sensory Organization Tests were evaluated with this system (Biodex Medical Systems, 2009). MSOT assesses the effects of somatosensory, visual and vestibular senses on postural control during the standing position. It evaluates the sensory component of balance in two different visual conditions and on two different support surfaces; condition 1: eyes open-firm surface, condition 2: eyes closed-firm surface, condition 3: eyes open-foam surface and condition 4: eyes closed-foam surface. Stability index scores were obtained as the test result

CONTACTS AND LOCATIONS:
Overall Officials: Taskin Ozkan, postgraduate, Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation Etlik, Ankara, Turkey, 06010, Ankara, Turkey (Türkiye)